CLINICAL TRIAL: NCT01808911
Title: Outcome of Acquired Haemophilia With Steroid Combined With Cyclophosphamide Versus Steroid Combined With Rituximab (CREHA Study)
Acronym: CREHA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 2011/090/HP
Record Dates: First submitted 2012-10-16; First posted 2013-03-11 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2025-09

CONDITIONS: Acquired Haemophilia
Keywords: Acquired haemophilia; Comparative and randomized study; Cyclophosphamide; Rituximab
MeSH Terms: interventions — Steroids; Cyclophosphamide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bras A (Active Comparator): Steroid 1mg/kg/d and Cyclophosphamide 2mg/kg/d
  Interventions: Drug: Steroid + cyclophosphamide
- Bras B (Experimental): Steroid 1mg/kg/d and Rituximab 375 mg/m2 every week during four weeks
  Interventions: Drug: Steroid + rituximab

INTERVENTIONS:
Drug: Steroid + cyclophosphamide
  Arms: Bras A
Drug: Steroid + rituximab
  Arms: Bras B

SUMMARY:
CREHA project is a study comparing steroid combined with cyclophosphamide versus steroid combined with rituximab in patients with acquired haemophilia. The study will test the hypothesis that steroid combined with cyclophosphamide is more effective than steroid plus rituximab for FVIII inhibitor eradication in acquired haemophilia.

DETAILED DESCRIPTION:
CREHA project is a multicenter, randomized, controlled efficacity and safety study comparing steroid combined with cyclophosphamide versus steroid combined with rituximab in patients with acquired haemophilia. The study will test the hypothesis that steroid combined with cyclophosphamide is more effective than steroid plus rituximab for FVIII inhibitor eradication in acquired haemophilia

ELIGIBILITY:
Inclusion Criteria:

* men or women
* women post-menpausal or with ongoing contraception
* 18 years old or more
* diagnosis of acquired hemophilia
* patient must be insured
* patient has provided written informed consent prior to enrolment
* patient compliant

Exclusion Criteria:

* constitutional hemophilia
* chemotherapy
* ongoing treatment with prednisone > 20mg further more 1 month
* ongoing treatment with prednisone >0.7 mg/d further more 10 days
* thrombocytopenia
* leukopenia
* chronic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2021-01-14 (Actual)

PRIMARY OUTCOMES:
Primary objective | During 18 months
  Demonstrate the inferiority of steroid combined with rituximab as compared to the recommended immunosuppressive approach (steroid combined with cysclophosphamide for 21 to 42 days) as the first-line immunosuppressive therapy for FVIII inhibitor eradication in acquired haemophilia
Primary efficacy outcome | During 18 months
  The primary efficacy outcome is the proportion of patients achieving complete remission defined as titer FVII inhibitor lower than 0.4 Bethesda unit and factor VIII level > 50%
Primary safety outcomes | During 18 months
  The primary safety outcomes will be the occurrence of major bleeding and infection related immunosuppressive treatment adverse events.

SECONDARY OUTCOMES:
Secondary objective | 6 months, 12 months and 18 months
  Secondary objective are time to complete remission, number of relapse at M6, M12, M18, adverse events (especially related to bleeding or to immunosuppressive treatment) and mortality
Other key safety outcome | During 18 months
  The other key safety outcome are clinically relevant non major bleeding, diabetes and mortality non-related with acquired haemophilia or immunosuppressive therapy

CONTACTS AND LOCATIONS:
Locations (34):
- France (34):
  - University Hospital Amiens, Amiens
  - Hospital of Béziers, Béziers
  - Hospital Jean Verdier, Bondy
  - Hospital Ambroise Paré, Boulogne-Billancourt
  - University Hospital of Brest - Hospital La cavale Blanche, Brest
  - University Hospital Côte de Nacre, Caen
  - University Hospital G. Montpied, Clermont-Ferrand
  - Hospital Henri Mondor, Créteil
  - University Hospital of Dijon - Hospital Général, Dijon
  - University Hospital Bocage, Dijon
  - University Hospital Michallon, Grenoble
  - Hospital Kremlin-Bicêtre, Le Kremlin-Bicêtre
  - University Regional Hospital of Lille, Lille
  - university Hospital of Limoges, Limoges
  - AP-HM, University Hospital La Conception, Marseille
  - University Hospital Saint-Eloi, Montpellier
  - Regional Center of Haemophilia Treatment (CRTH) de Lorraine, Nancy
  - University Hospital of Nantes, Hospital Hôtel-Dieu, Nantes
  - Hospital Archet 1, Nice
  - Hospital Bichat, Paris
  - Hospital Saint-Louis, Paris
  - Hospital Pitié-Salpêtrière, Paris
  - Hospital Cochin, Paris
  - Europen Hospital of Georges Pompidou (HEGP), Paris
  - University Hospital of Bordeaux - Hospital Haut-Lévêque, Pessac
  - Hospital Lyon Sud, Pierre-Bénite
  - University Hospital of Poitiers, Poitiers
  - Hospital Sud / Hospital Pontchaillou, Rennes
  - University Hospital of Rouen, Rouen
  - Hospital Nord, Saint-Etienne
  - University Regional Hospital Hautepierre, Strasbourg
  - Hospital Purpan, Toulouse
  - Hospital Rangueil, Toulouse
  - Hopsital Bretonneau, Tours

REFERENCES:
- [Derived] Levesque H, Viallard JF, Houivet E, Bonnotte B, Voisin S, Le Cam-Duchez V, Maillot F, Lambert M, Liozon E, Hervier B, Fain O, Guillet B, Schmidt J, Luca LE, Ebbo M, Ferreira-Maldent N, Babuty A, Sailler L, Duffau P, Barbay V, Audia S, Benichou J, Graveleau J, Benhamou Y; CREHA Study investigators on behalf the scientific committee of the "Societe Nationale Francaise de Medecine Interne" (SNFMI - French National Society of Internal Medicine). Cyclophosphamide vs rituximab for eradicating inhibitors in acquired hemophilia A: A randomized trial in 108 patients. Thromb Res. 2024 May;237:79-87. doi: 10.1016/j.thromres.2024.03.012. Epub 2024 Mar 15. PMID 38555718